CLINICAL TRIAL: NCT07084402
Title: Short-term Bactericidal Effect of Contezolid in Mycobacterium Avium Complex Pulmonary Disease
Brief Title: Short-term Bactericidal Effect of Contezolid in MAC-PD
Acronym: CONTE-MAC
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Bin Cao (Other)
Collaborators: Beijing Chest Hospital, Capital Medical University (Other); Jiangxi Provincial Chest Hospital (Unknown); MicuRx (Industry)
Responsible Party: Sponsor-Investigator, Bin Cao, Professor, Capital Medical University
Organization: Capital Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-HX-59
Record Dates: First submitted 2025-07-17; First posted 2025-07-24 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Mycobacterium Avium Complex Pulmonary Disease
MeSH Terms: interventions — contezolid; Rifampin; Ethambutol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Contezolid plus standard regimen (Experimental): Participants in this arm will receive contezolid 800mg po q12h, azithromycin 500mg po tiw (250mg po tiw if weight below 50kg), rifampicin 600mg po tiw and ethambutol 25mg/kg po tiw for 6 months.
  Interventions: Drug: Contezolid; Drug: Azithromcyin; Drug: Rifampicin (RIF); Drug: Ethambutol
- Standard regimen (Active Comparator): Participants in this arm will receive azithromycin 500mg po tiw (250mg po tiw if weight below 50kg), rifampicin 600mg po tiw and ethambutol 25mg/kg po tiw for 6 months.
  Interventions: Drug: Azithromcyin; Drug: Rifampicin (RIF); Drug: Ethambutol

INTERVENTIONS:
Drug: Contezolid — contezolid 800mg po q12h for 6 months
  Arms: Contezolid plus standard regimen
Drug: Azithromcyin — azithromycin 500mg po tiw (250mg po tiw if weight below 50kg) for 6 months.
Drug: Rifampicin (RIF) — rifampicin 600mg po tiw for 6 months.
Drug: Ethambutol — ethambutol 25mg/kg po tiw for 6 months.

SUMMARY:
The goal of this clinical trial is to learn if contezolid works to treat mycobacterium avium complex pulmonary disease in adults. It will also learn about the safety of contezolid. The main questions it aims to answer are:

Does adding contezolid to standard regimen further decrease the bacterial load in patients' sputum compared with current standard regimen? What medical problems do participants have when taking contezolid along with standard regimen? Researchers will compare standard regimen plus contezolid to standard regimen alone to see if contezolid helps further lower the count of bacteria in patients' sputum.

Participants will:

Take contezolid and standard regimen (azithromycin, ethambutol and rifampicin) or standard regimen only for 6 months, contezolid is administered every day while other drugs are taken 3 times a week Visit the clinic once every 1 month for checkups and tests.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily participate in this study and sign the Informed Consent Form.
2. Age ≥ 18 years and ≤75 years; gender unrestricted.
3. Confirmed diagnosis of MAC pulmonary disease per ATS/IDSA 2020 guidelines or Chinese Guidelines for Diagnosis and Treatment of Nontuberculous Mycobacterial Diseases (2020 edition), with imaging features consistent with nodular bronchiectatic type.
4. No prior anti-MAC treatment within the 3 months preceding screening.
5. For premenopausal women of childbearing potential who are not surgically sterile:

   Must use a medically accepted contraceptive method (e.g., intrauterine device, hormonal contraception, or condom) during the study period and for 3 months following the last dose of investigational treatment.

   Serum or urine human chorionic gonadotropin (hCG) test must be negative within 72 hours prior to enrollment.

   Must not be breastfeeding. Male patients with partners of childbearing potential must use effective contraception during the study period and for 3 months after the last dose.
6. Organ function criteria met within one week prior to enrollment:

i. Hemoglobin ≥60 g/L; ii. Neutrophil count ≥0.5 × 10⁹/L; iii. Platelet count ≥60 × 10⁹/L; iv. Serum total bilirubin ≤3 × upper limit of normal (ULN); v. Aspartate aminotransferase (AST) ≤3 × ULN; vi. Alanine aminotransferase (ALT) ≤3 × ULN; vii. Serum creatinine <2 × ULN OR creatinine clearance ≥60 mL/min; viii. Blood urea nitrogen (BUN) ≤200 mg/L; ix. Urinalysis: Proteinuria <++; if proteinuria is +, 24-hour total protein must be <500 mg.

x. Fasting blood glucose within normal range OR stable glycemic control in diabetic patients.

xi. Cardiac function: No myocardial infarction in the preceding 6 months; No unstable angina or severe arrhythmias; New York Heart Association (NYHA) functional class >II.

Exclusion Criteria:

1. History of allergy to any study drug in the treatment regimen.
2. Mixed infections with multiple mycobacteria, bacteria, fungi, or viruses (e.g., HIV coinfection).
3. Presence of congenital/acquired immunodeficiency disorders, active pulmonary malignancy (primary or metastatic), or other malignancies requiring chemotherapy/radiation therapy during the screening or study period.
4. History of solid organ transplantation.
5. Currently undergoing dialysis.
6. Uncontrolled radiation pneumonitis requiring steroid or immunoglobulin pulse therapy, active interstitial lung disease with clinical evidence, uncontrolled and significant pleural effusion or pericardial effusion.
7. Unstable systemic comorbidities including:

   Hypertensive crisis; Unstable angina; Congestive heart failure (NYHA Class III/IV); Myocardial infarction within the preceding 6 months; Severe psychiatric disorders requiring medication (e.g., schizophrenia, bipolar disorder); Severe hepatic or renal dysfunction (e.g., Child-Pugh Class C cirrhosis, eGFR <30 mL/min/1.73m²); Neurodegenerative diseases (e.g., Alzheimer's disease).
8. Poor gastrointestinal function or malabsorption syndrome.
9. Receipt of other investigational drugs within 4 weeks prior to the first study drug administration.
10. Concurrent participation in another interventional clinical trial, unless it is an observational/noninterventional study OR follow-up phase of a completed intervention trial.
11. Any physical examination findings or clinical tests deemed by the investigator as likely to:

Interfere with study results; Increase risks of complications during treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2025-07-24 (Actual); Primary Completion 2027-07-24 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
time-to-positivity of sputum mycobacterium culture | the end of month 3

SECONDARY OUTCOMES:
culture conversion | at the end of month 3 and 6
time to first culture conversion | from enrollment to the end of month 6
CT status of the lesion | at the end of month 3 and 6
adverse events | from enrollment to the end of month 6

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojing Cui, M.D., Principal Investigator — China-Japan Friendship Hospital
Locations (3):
- China (3):
  - Beijing Chest Hospital, Capital Medical University, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Jiangxi Provincial Chest Hospital, Nanchang, Jiangxi

IPD SHARING:
Plan to Share IPD: No